CLINICAL TRIAL: NCT01999764
Title: Evaluation of the Effects of Oral QLT091001 in Adults With Impaired Dark Adaptation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: QLT Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RET IDA 02
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-06

CONDITIONS: Impaired Dark Adaptation
MeSH Terms: interventions — retinol acetate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (for QLT091001) (Placebo Comparator): Placebo is supplied to mimic QLT091001 oral solution.
  Interventions: Other: Placebo
- QLT091001 - first oral dose (Experimental): Subjects will receive an oral dose of 10mg/m2 of QLT091001.
  Interventions: Drug: QLT091001
- QLT091001 - second oral dose (Experimental): Subjects will receive an oral dose of 40 mg/m2 of QLT091001.
  Interventions: Drug: QLT091001

INTERVENTIONS:
Drug: QLT091001 — QLT091001 administered orally at multiple time points.
  Arms: QLT091001 - first oral dose; QLT091001 - second oral dose
Other: Placebo — Placebo is administered orally at multiple time points.
  Arms: Placebo (for QLT091001)

SUMMARY:
This is a Phase IIa proof-of-concept study to evaluate the effects of oral QLT091001 on adults with impaired dark adaptation.

DETAILED DESCRIPTION:
This proof-of-concept study is a randomized, parallel design of two different oral doses of QLT091001 compared to placebo to evaluate treatment effects in patients with impaired dark adaptation.

Approximately 40 subjects will be enrolled in this study at approximately 7 centers in the US.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥60 yrs with early age-related macular degeneration (AMD) based on LLLC BCVA criterion or evidence of impaired dark adaptation
* Subjects with high luminance high contrast best-corrected visual acuity (HLHC BCVA) of 40 letters (20/40 Snellen) or better in the study eye
* Capable and willing to provide consent

Exclusion Criteria:

* Women of child bearing potential
* Subjects with late AMD or any other optic neuropathy in the study eye
* Subjects with posterior subcapsular cataract or multifocal intra-ocular lens (IOL) in the study eye
* Subjects who are actively participating in an experimental therapy study or who have received experimental therapy within 60 days of Day 0 or who have taken any prescription/investigational oral retinoid medication within 6 months of Day 0
* Subjects taking age-related eye disease study (AREDS) supplements containing beta-carotene

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | Through 7 weeks
  Low luminance low contrast best-corrected visual acuity (LLLC BCVA) will be measured at multiple time points.

SECONDARY OUTCOMES:
Dark Adaptation Time | Through 7 weeks
  Dark Adaptation Time will be measured at multiple time points.

OTHER OUTCOMES:
Glare Recovery | Through 7 weeks
  Glare recovery time will be measured at multiple time points.

CONTACTS AND LOCATIONS:
Overall Officials: Sushanta Mallick, Ph.D MBA, Study Director — QLT Inc.
Locations (7):
- United States (7):
  - Sall Research Medical Center, Artesia, California
  - California Retina Consultants, Santa Barbara, California
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Keystone Research Ltd., Austin, Texas
  - Retina Foundation of the Southwest, Dallas, Texas
  - Retina Consultants of Houston, Houston, Texas
  - Proliance Surgeons Inc., Seattle, Washington